CLINICAL TRIAL: NCT03871075
Title: Intermittent Pneumatic Compression With and Without Exercise to Improve Functioning in Peripheral Artery Disease: The INTERCEDE TRIAL
Brief Title: Intermittent Pneumatic Compression With and Without Exercise to Improve Functioning in Peripheral Artery Disease
Acronym: INTERCEDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00208245; 1R01AG057693-01A1 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-03-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral arterial disease; Peripheral Artery Disease; PAD; exercise; Intermittent claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity; Intermittent Claudication | interventions — Intermittent Pneumatic Compression Devices; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Group assignment regarding the intermittent pneumatic compression device is double-blinded and neither investigators nor participants in the study will know which intermittent pneumatic compression device each participant has (therapeutic intervention vs. sham). Participants will be aware of their exercise group assignment after randomization, but the study coordinators collecting follow-up data will be unaware of each participant's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- IPC + exercise (Experimental): Participants will be asked to wear the intermittent pneumatic compression device for up to three hours daily. They will be helped to engage in home-based walking exercise therapy.
  Interventions: Device: intermittent pneumatic compression; Behavioral: exercise
- IPC + "no exercise" control (Experimental): Participants will be asked to wear the intermittent pneumatic compression device for up to three hours daily. They will be asked to participate in an educational/informational intervention consisting of an attention control intervention
  Interventions: Device: intermittent pneumatic compression; Behavioral: Health Education
- sham control + exercise (Active Comparator): Participants will be asked to wear a sham intermittent pneumatic compression device for up to three hours daily. The sham device inflates at the same frequency, but to a much lower systolic pressure, compared to the therapeutic pneumatic compression device. Participants in this group will be helped to engage in home-based walking exercise therapy.
  Interventions: Behavioral: exercise; Device: Sham device
- sham control + "no exercise" control (Active Comparator): Participants will be asked to wear a sham intermittent pneumatic compression device for up to three hours daily. The sham device inflates at the same frequency, but to a much lower systolic pressure, compared to the therapeutic pneumatic compression device. Participants will be asked to participate in an educational/informational intervention, designed as an attention control group.
  Interventions: Device: Sham device; Behavioral: Health Education

INTERVENTIONS:
Device: intermittent pneumatic compression — Intermittent pneumatic compression is a non-invasive intervention, consisting of an air pump inside inflatable cuffs that are wrapped around the feet, ankles, and calves. The cuffs rapidly inflate to a pressure of 120 mm Hg, which is sustained for three seconds, followed by rapid deflation. Participants will be asked to wear the device for two hours daily. The device will inflate 180 times/hour.
  Other Names: IPC
  Arms: IPC + "no exercise" control; IPC + exercise
Behavioral: exercise — Participants will be asked to walk for exercise five days/week, working up to 50 minutes of exercise per day. The intervention includes a) group meetings at the medical center with the coach and other PAD participants; b) regularly scheduled individual telephone check-in by the coach c) weekly remote monitoring by the coach; d) use of the activity monitor to monitor exercise intensity and duration.
  Arms: IPC + exercise; sham control + exercise
Device: Sham device — The sham control device is a non-invasive intervention, consisting of an air pump inside inflatable cuffs that are wrapped around the feet, ankles, and calves. The cuffs rapidly inflate to a pressure of 25 mm Hg, which is sustained for three seconds, followed by rapid deflation. Participants will be asked to wear the device for two hours daily. The device will inflate 180 times/hour.
  Arms: sham control + "no exercise" control; sham control + exercise
Behavioral: Health Education — Participants attend health-education lectures and receive telephone calls at the same frequency as the exercise group. On-site lectures are delivered by faculty and staff at the medical center. Telephone calls review health-related handouts from the NIA website that are mailed in advance of the telephone call. Content does not include exercise information.
  Arms: IPC + "no exercise" control; sham control + "no exercise" control

SUMMARY:
The INTERCEDE randomized trial will establish whether six-months of intermittent pneumatic compression combined with walking exercise improves walking endurance at six-month follow-up, compared to walking exercise + sham compression therapy, in people with lower extremity peripheral artery disease (PAD). The INTERCEDE trial will also determine whether intermittent pneumatic compression therapy improves walking endurance at 6-month follow-up, compared to a sham compression therapy. The trial will also determine whether benefits of intermittent pneumatic compression persist after intermittent pneumatic compression treatment is completed.

DETAILED DESCRIPTION:
Walking exercise is first-line therapy for PAD. However, many PAD patients are unable or unwilling to exercise. Therefore, in people with PAD, the investigators will determine whether intermittent pneumatic compression augments the benefits of exercise and whether intermittent pneumatic compression alone improves walking performance compared to sham control. The investigators will conduct a randomized trial (2 x 2 factorial design) of 230 PAD participants randomized to one of four groups: Group A: intermittent pneumatic compression + exercise; Group B: intermittent pneumatic compression+ "no exercise" control; Group C: sham control + exercise; and Group D: sham control + "no exercise" control. The intermittent pneumatic compression and sham interventions will be delivered for six months. The primary outcome is change in six-minute walk distance at 6-month follow-up. In secondary aims, the investigators will determine whether the benefits of intermittent pneumatic compression persist even after intermittent pneumatic compression is discontinued and delineate mechanisms by which intermittent pneumatic compression affects walking performance, by measuring changes in MRI-measured calf muscle perfusion and physical activity. The investigators will determine whether intermittent pneumatic compression improves systemic endothelial function, by measuring changes in brachial artery flow-mediated dilation (FMD).

ELIGIBILITY:
Inclusion Criteria:

All participants will have PAD. PAD will be defined as follows: first, an ankle-brachial index (ABI) < or = 0.90 at the baseline study visit is an inclusion criterion for PAD. Second, potential participants with an ABI >0.90 who have vascular laboratory evidence of PAD. Vascular laboratory evidence consists of objective evidence of PAD, including toe brachial index (TBI) < or = 0.70, Duplex measure showing 70% stenosis or greater, or ABI values < 0.90. Abnormal waveforms or pulse volume recordings alone from a non-invasive vascular laboratory test will not be sufficient for enrollment. Third, potential participants with an ABI >0.90 who have angiographic evidence of PAD consisting of a stenosis of 70% or greater in a lower extremity artery.

Exclusion Criteria:

1. Above- or below-knee amputation.
2. Critical limb ischemia or ABI < 0.30 in the setting of ischemic symptoms at rest or physical examination findings consistent with critical limb ischemia. Some potential participants with symptoms or signs of critical limb ischemia may be excluded at the principal investigator's discretion if the ABI is 0.30 or higher.
3. Wheelchair-bound.
4. Current foot ulcer on bottom of foot.
5. Walking is primarily limited by a symptom other than PAD.
6. Failure to successfully complete the study run-in.
7. Major surgery, revascularization, or orthopedic surgery in the past 3 months or planned in the next 12 months.
8. Major medical illness including Parkinson's Disease, lung disease requiring oxygen, cancer requiring treatment in the previous two years, or life-threatening illness with a life expectancy of less than six months. Participants who only use oxygen at night will be potentially eligible. [NOTE: potential participants treated for cancer in the past two years may still qualify if they have had treatment for early stage cancer in the past two years and the prognosis is excellent. Potential participants treated for basal cell or squamous cell skin cancer will not be excluded.]
9. Already exercising at a level consistent with exercise intervention. Current or recent participation in exercise rehabilitation (within the past three months).
10. Recently diagnosed (within the past three months) with acute lower extremity deep venous thrombosis, pulmonary embolism, or severe heart failure (i.e. New York Heart Association (NYHA) Class III or IV).
11. Mini-Mental Status Examination (MMSE) score <23 or dementia.
12. Participation in or completion of a clinical trial in the previous three months.
13. Non-English speaking.
14. Increase in angina in the past month, angina at rest, or abnormal baseline treadmill stress test. Potential participants may become eligible after an abnormal baseline treadmill stress test if they have evidence of an absence of coronary ischemia based on testing (such as a stress test with imaging or a coronary angiogram) from a test performed with their own physician and if they do not have symptoms of unstable angina. The evidence of absent coronary ischemia, based on an imaging stress test or coronary angiogram, must have been performed within the previous year.
15. Ongoing infection of the toes, foot, or lower extremity.
16. Potential participants who started on cilostazol within the last three months. They may be evaluated for eligibility once three months have passed since beginning cilostazol.
17. Significant peripheral edema, defined as 3+ or greater edema severity, as determined by the principal investigator.
18. BMI >45 kg/M2
19. Significant visual impairment that interferes with walking.
20. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk distance (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression combined with exercise improves the 6-minute walk at 6-month follow-up compared to exercise alone.
Six-minute walk distance (intermittent pneumatic compression therapy alone (without exercise) vs. sham alone (without exercise) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone (without exercise) improves the 6-minute walk at 6-month follow-up, compared to the sham control alone (without exercise).

SECONDARY OUTCOMES:
Six-minute walk distance (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves the six-minute walk at 12-month follow-up, 6 months after the intermittent pneumatic compression therapy intervention is completed, compared to exercise alone.
Six-minute walk distance (IPC only v. sham only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves the six-minute walk distance at 12-month follow-up, 6 months after the intermittent pneumatic compression therapy intervention is completed, compared to the sham control.
Calf muscle perfusion (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves calf muscle perfusion at 6-month follow-up, compared to exercise alone.
Brachial artery FMD (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves brachial artery FMD at 6-month follow-up, compared to exercise alone.
Physical Activity measured by Actigraph activity monitor (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves physical activity measured by Actigraph activity monitor at 6-month follow-up, compared to exercise alone.
Calf muscle perfusion (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves calf muscle perfusion at 12-month follow-up, compared to exercise alone.
Brachial artery FMD (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves brachial artery FMD at 12-month follow-up, compared to exercise alone.
Physical Activity measured by Actigraph activity monitor (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves physical activity measured by Actigraph activity monitor at 12-month follow-up, compared to exercise alone.
Calf muscle perfusion (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves calf muscle perfusion at 6-month follow-up, compared to the sham control.
Brachial artery FMD (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves brachial artery FMD at 6-month follow-up, compared to the sham control.
Physical Activity measured by Actigraph activity monitor (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves physical activity measured by Actigraph activity monitor at 6-month follow-up, compared to the sham control.
Calf muscle perfusion (intermittent pneumatic compression therapy only v. sham only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves calf muscle perfusion at 12-month follow-up, compared to the sham control.
Brachial artery FMD (intermittent pneumatic compression therapy only v. sham only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves brachial artery FMD at 12-month follow-up, compared to the sham control.
Physical Activity measured by Actigraph activity monitor (intermittent pneumatic compression therapy only v. sham only) | Baseline to 12-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves physical activity measured by Actigraph activity monitor at 12-month follow-up, compared to the sham control.

OTHER OUTCOMES:
Mitochondrial biogenesis (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves mitochondrial biogenesis (PGC-1α) at 6-month follow- up, compared to exercise alone.
Mitochondrial activity (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves mitochondrial activity (Cytochrome C oxidase) at 6-month follow- up, compared to exercise alone.
Vascular endothelial growth factor abundance (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves vascular endothelial growth factor abundance at 6-month follow- up, compared to exercise alone.
Anti-oxidant enzyme activity (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves anti-oxidant enzyme activity (MnSOD) at 6-month follow- up, compared to exercise alone.
Immunohistochemistry-measured mitochondrial activity (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves immunohistochemistry-measured mitochondrial activity (COX and SDH) at 6-month follow- up, compared to exercise alone.
Autophagy (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves autophagy (LC3, LAMP2, PARKIN) at 6-month follow- up, compared to exercise alone.
Capillary density (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves capillary density (CD31) at 6-month follow- up, compared to exercise alone.
Satellite cell content (intermittent pneumatic compression therapy + exercise v. exercise only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy combined with exercise improves satellite cell content (Pax7) at 6-month follow- up, compared to exercise alone.
Mitochondrial biogenesis (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves mitochondrial biogenesis (PGC-1α) at 6-month follow- up, compared to the sham control.
Mitochondrial activity (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves mitochondrial activity (Cytochrome C oxidase) at 6-month follow- up, compared to the sham control.
Vascular endothelial growth factor abundance (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves vascular endothelial growth factor abundance at 6-month follow- up, compared to the sham control.
Anti-oxidant enzyme activity (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves anti-oxidant enzyme activity (MnSOD) at 6-month follow- up, compared to the sham control.
Immunohistochemistry-measured mitochondrial activity (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves immunohistochemistry-measured mitochondrial activity (COX and SDH) at 6-month follow- up, compared to the sham control.
Autophagy (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves autophagy (LC3, LAMP2, PARKIN) at 6-month follow- up, compared to the sham control.
Capillary density (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves capillary density (CD31) at 6-month follow- up, compared to the sham control.
Satellite cell content (intermittent pneumatic compression therapy only v. sham only) | Baseline to 6-month follow-up
  Among PAD participants, the investigators will determine whether intermittent pneumatic compression therapy alone improves satellite cell content (Pax7) at 6-month follow- up, compared to the sham control

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern Universtiy
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Nayak P, Polonsky T, Tian L, Greenland P, Xu S, Zhang D, Zhao L, Criqui MH, Kibbe MR, Gladders B, Goodney P, Ho K, Guralnik JM, McDermott MM. Medical therapies, comorbid conditions, and functional performance in people with peripheral artery disease enrolled in clinical trials between 2004 and 2021. Vasc Med. 2023 Apr;28(2):144-146. doi: 10.1177/1358863X221145533. Epub 2023 Jan 1. PMID 36588397